CLINICAL TRIAL: NCT03635034
Title: Examining the Routine Use of Bladder Catheters During Atrial Fibrillation Procedures
Brief Title: Bladder Catheters During Ablation Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Vincent Cardiovascular Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R20180053
Record Dates: First submitted 2018-07-27; First posted 2018-08-17 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Atrial Fibrillation; Catheter Ablation; Catheter Complications
Keywords: urinary catheter; catheter ablation procedures
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: We will compare the two groups for complications related to catheter or not having a catheter placed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- No Bladder catheter (Experimental): Subjects will not have bladder catheter inserted during their ablation procedure.
  Intervention: No catheter
  Interventions: Device: No catheter
- Bladder catheter inserted (Active Comparator): Bladder catheter will be inserted prior to starting ablation procedure after the subject is under general anesthesia.
  Intervention: bladder catheter inserted
  Interventions: Device: Insert bladder catheter

INTERVENTIONS:
Device: Insert bladder catheter — Bladder catheter will be inserted according to randomization schema
  Arms: Bladder catheter inserted
Device: No catheter — Subjects will not receive a bladder catheter during the ablation procedure
  Arms: No Bladder catheter

SUMMARY:
Inserting a Bladder catheter during catheter ablation is standard practice at most Institutions. Unfortunately, bladder catheters are associated with adverse outcomes, including catheter associated cystitis, hematuria, dysuria, and urethral damage.

The investigator proposes a prospective, randomized clinical trial comparing group A that will receive a catheter during the ablation procedure and group B that will not receive the procedure. The Investigator hypothesizes the group receiving the bladder catheters will have a higher rate of complications.

DETAILED DESCRIPTION:
(AF) is the commonest arrhythmia worldwide and accounts for significant morbidity. The mainstay of treatment for drug refractory AF is catheter ablation. A preponderance of evidence indicates better outcomes when this procedure is performed under general anesthesia; this is standard of care at our institution. However, for a variety of reasons including long procedure time, procedural intravenous fluid administration, and prolonged bedrest following the procedure, standard of care at our institution and others is for bladder catheter placement during the procedure (4). Unfortunately, bladder catheters used during cardiac surgery have been associated with adverse outcomes, including catheter associated cystitis, hematuria, dysuria, and urethral damage(

Fortunately, the landscape of AF ablation is changing rapidly, and procedure times are rapidly decreasing. Improvements in three dimensional mapping technology has allowed for less reliance on fluoroscopy and allows for real time visualization of ablation lesions. Improvements in ablation catheters have allowed for significantly reduced intravenous fluid administration during the procedure. The Site has also adopted an expedited protocol for venous hemostasis following the procedure that involves a figure-of-eight groin stitch, allowing for earlier mobility and a shorter bed rest following the procedure. Therefore, we question the need for routine bladder catheter placement during AF ablation procedures

ELIGIBILITY:
Inclusion Criteria:

* All subjects presenting to the St. Vincent EP lab for AF ablation Ability to sign informed consent

Exclusion Criteria:

* Recent (within 1 month) cystitis, history of urinary retention or incontinence, prior bladder catheter associated complications, hematuria, chronic kidney disease (stage II, III, IV, or V), dialysis, prostate cancer, renal cancer, bladder cancer, expected procedure duration >6 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2020-01-16 (Actual)

PRIMARY OUTCOMES:
Composite of catheter associated complications at day one and thirty will be assessed among the two arms - those with bladder catheters and those who did not receive the bladder catheter during the ablation procedure. | Post-op day 1 and 30 days
  Per patient reported outcomes, subjects will be asked if they experienced any of the following complications: cystitis, hematuria, dysuria, urethral damage and urinary retention. The primary composite outcome of cystitis, hematuria, dysuria, urethral damage or urinary retention will be compared using Chisq or Fisher's exact test. Additional bivariate correlates to the primary outcome will be analysed including age, gender, operator, procedure satisfaction score, procedure duration, procedural fluid administration, total hospital stay fluid administration, and baseline clinical variables. Variables with p value <o.o5 on bivariate analysis will be included in a multivariate regression model.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Vincent Hospital and Healthcare Center, Indianapolis, Indiana, United States